CLINICAL TRIAL: NCT03483246
Title: Impact of Fecal Microbiota Transplantation in Ulcerative Colitis: a Randomized, Sham Controlled Trial
Brief Title: Impact of Fecal Microbiota Transplantation in Ulcerative Colitis
Acronym: REBALANCE-UC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CRB-HUEP (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P 160931J; 2017-003802-42 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Inflammatory bowel disease; Fecal microbiota transplantation
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B - fecal microbiota transplantation (Experimental): Patients receiving the fecal microbiota transplantation (FMT) in 3 times after inclusion and randomisation
  Interventions: Drug: Fecal Microbiota Transplantation (FMT)
- Group A- Sham-transplantation (Placebo Comparator): Patients receiving the sham-transplantation in 3 times after inclusion and randomisation
  Interventions: Drug: Sham-transplantation Placebo

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation (FMT) — The colonoscopy for FMT will be planned as soon as possible and never more than 5 weeks after inclusion visit.
  After colon cleansing using Polyethylen glycol, the patient will have a colonoscopy under general anesthesia.
  The patient will then receive either FMT (frozen preparation of 50g of stools in 300ml of physio, see donor section for details) or sham transplantation (FMT vehicle) in the cecum.
  Arms: Group B - fecal microbiota transplantation
Drug: Sham-transplantation Placebo — The sham-transplantation will be planned as soon as possible and never more than 5 weeks after inclusion visit.
  After colon cleansing using Polyethylen glycol, the patient will have a colonoscopy under general anesthesia.
  The patient will then sham transplantation (FMT vehicle) in the cecum.
  Arms: Group A- Sham-transplantation

SUMMARY:
Ulcerative colitis (UC) is a chronic relapsing inflammatory bowel disease. UC pathogenesis remains poorly understood but involves an inappropriate immune response toward an unbalanced gut microbiota (called dysbiosis) in predisposed hosts.

The purpose of this study is to determine the effect of the fecal microbiota transplantation on UC.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic relapsing inflammatory bowel disease affecting approximately 90 000 patients in France, mostly at young age, and altering their quality of life.

Conventional Immunosuppressive treatment (ie azathioprine, anti-TNF (tumor necrosis factor ), vedolizumab) used in UC are expensive and associated with potentially severe complications such as infections and cancers.

UC pathogenesis remains poorly understood but involves an inappropriate immune response toward an unbalanced gut microbiota (called dysbiosis) in predisposed hosts.

Fecal microbiota transplantation (FMT) is now recommended in guidelines for treating recurrent Clostridium difficile infection. Although the pathogenesis involved in UC is different, FMT is a potential therapeutic strategy as transferring a healthy microbiota in an UC patient could restore the appropriate host-microbiota crosstalk.

As the gut microbiota is dramatically altered by intestinal inflammation, transferring a massive amount of microbial organisms in an inflamed gut with epithelial barrier disruption might be a suboptimal strategy and could even have detrimental effects by allowing bacterial translocation.

Thus, it's possible that performing FMT in UC patients who achieved remission after conventional treatment might be associated with better clinical outcome than in patients with active disease.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for patients :

* Age ≥ 18 years and < 75 years
* Ulcerative colitis (according to the Lennard Jones criteria) diagnosed for at least 3 months and :

  * Currently active (PMC > 1) and planned to be treated by systemic corticosteroids (minimum 40mg prednisone equivalent daily) Or
  * Currently treated by systemic corticosteroid (minimum 40 mg prednisone equivalent daily) within max 3 weeks Or
  * Steroid dependent patients (at least one unsuccessful attempt to discontinue steroid within the last 6 months before inclusion)
* Patient with health insurance (AME excepted)
* Informed written consent
* Female of child-bearing age with an active contraception and this during at least period of treatment until the end of active follow-up period (week 24)

Inclusion Criteria for healthy volunteers donors :

* Age ≥ 18 years and < 50 years
* 17 kg/m² < body mass index < 30 kg/m²
* Regular bowel movement defined as at least 1 stool every other day and maximum 2 stools per day
* Subject with health insurance (AME excepted)
* Informed Written consent

Exclusion Criteria:

Exclusion Criteria for patients :

* UC complication requiring surgical treatment
* Patient treated with high dose corticosteroid more than three weeks before inclusion (≥ 40 mg prednisone equivalent daily) except in case of steroid-dependence
* Contraindication to colonoscopy or anesthesia
* Pregnancy or breastfeeding during the study
* Treatment preceding the colonoscopy with:

  * intravenous infliximab and/or vedolizumab and/or ustekinumab (< 6 weeks before the planned date of the colonoscopy) and/or subcutaneous infliximab (<2 weeks before the planned date of the colonoscopy), and /or adalimumab (<2 weeks before the planned date of the colonoscopy) and/or golimumab and/or tofacitinib (<4 weeks before the planned date of the colonoscopy)
  * immunosuppressant (thiopurine, methotrexate, tacrolimus or other classical immunosuppressant) started or stopped < 3 months before the planned date of the colonoscopy
  * Antibiotics, antifungic or probiotics treatment < 4 weeks before the planned date of the colonoscopy
* participation in any other interventional study
* patient under legal protection

Exclusion Criteria for healthy volunteers donors :

- For details, please see protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Steroid-free clinical and endoscopic remission | 12 weeks after FMT or sham-transplantation
  Steroid-free clinical and endoscopic remission defined as a total Mayo score of 2 or lower and no subscore higher than 1 and mucosal healing defined as an endoscopic subscore of 0 or 1 (Sigmoidoscopy).

SECONDARY OUTCOMES:
Steroid-free clinical remission | 12 weeks after FMT or sham-transplantation
  Steroid-free clinical remission defined as a Partial Mayo Clinic score of 0 or 1
Steroid-free clinical remission | 24 weeks after FMT or sham-transplantation
  Steroid-free clinical remission defined as a Partial Mayo Clinic score of 0 or 1
Steroid-free endoscopic response | 12 weeks after FMTor sham-transplantation
  Steroid-free endoscopic response defined as a Mayo endoscopy subscore of 1 or less, with a reduction of at least 1 point from baseline
Steroid-free endoscopic remission | 12 weeks after FMT or sham-transplantation
  Steroid-free endoscopic remission defined as an Endoscopic Mayo Clinic score of 0
Microbiota composition and diversity | 12 and 24 weeks after FMT or sham-transplantation
  Microbiota composition and diversity assessed by 16s sequencing compared to baseline and to donor's microbiota.
Proportion of adverse events in each group | Through study completion, up to 25 months and one week
  abdominal pain, nausea, vomiting, fever, modified intestinal transit and episode of infection
Inflammatory biological parameter 1 | up to 24 weeks
  CRP
Inflammatory biological parameter 2 | up to 24 weeks
  fecal calprotectin
Inflammatory biological parameter 3 | up to 24 weeks
  platelet number
Endoscopic lesions | 12 weeks after FMT or sham-transplantation
  Endoscopic lesions at coloscopy and sigmoidoscopy by endoscopic Mayo score
Endoscopic lesions | 12 weeks after FMT or sham-transplantation
  Endoscopic lesions at coloscopy (baseline) and sigmoidoscopy by UCEIS score

CONTACTS AND LOCATIONS:
Overall Officials: Harry SOKOL, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Gastroentérologie et Nutrition Hôpital Saint Antoine, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ananthakrishnan AN. Epidemiology and risk factors for IBD. Nat Rev Gastroenterol Hepatol. 2015 Apr;12(4):205-17. doi: 10.1038/nrgastro.2015.34. Epub 2015 Mar 3. PMID 25732745
- [Background] Angelberger S, Reinisch W, Makristathis A, Lichtenberger C, Dejaco C, Papay P, Novacek G, Trauner M, Loy A, Berry D. Temporal bacterial community dynamics vary among ulcerative colitis patients after fecal microbiota transplantation. Am J Gastroenterol. 2013 Oct;108(10):1620-30. doi: 10.1038/ajg.2013.257. Epub 2013 Sep 24. PMID 24060759
- [Background] Beaugerie L, Itzkowitz SH. Cancers Complicating Inflammatory Bowel Disease. N Engl J Med. 2015 Jul 9;373(2):195. doi: 10.1056/NEJMc1505689. No abstract available. PMID 26154801
- [Background] Best WR, Becktel JM, Singleton JW, Kern F Jr. Development of a Crohn's disease activity index. National Cooperative Crohn's Disease Study. Gastroenterology. 1976 Mar;70(3):439-44. PMID 1248701
- [Background] Borody T, Fischer M, Mitchell S, Campbell J. Fecal microbiota transplantation in gastrointestinal disease: 2015 update and the road ahead. Expert Rev Gastroenterol Hepatol. 2015;9(11):1379-91. doi: 10.1586/17474124.2015.1086267. Epub 2015 Sep 28. PMID 26414076
- [Background] Colman RJ, Rubin DT. Fecal microbiota transplantation as therapy for inflammatory bowel disease: a systematic review and meta-analysis. J Crohns Colitis. 2014 Dec;8(12):1569-81. doi: 10.1016/j.crohns.2014.08.006. Epub 2014 Sep 13. PMID 25223604
- [Background] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735
- [Background] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601
- [Background] Grinspan AM, Kelly CR. Fecal Microbiota Transplantation for Ulcerative Colitis: Not Just Yet. Gastroenterology. 2015 Jul;149(1):15-8. doi: 10.1053/j.gastro.2015.05.030. Epub 2015 May 27. No abstract available. PMID 26021232
- [Background] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Khor B, Gardet A, Xavier RJ. Genetics and pathogenesis of inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):307-17. doi: 10.1038/nature10209. PMID 21677747
- [Background] Lamas B, Richard ML, Leducq V, Pham HP, Michel ML, Da Costa G, Bridonneau C, Jegou S, Hoffmann TW, Natividad JM, Brot L, Taleb S, Couturier-Maillard A, Nion-Larmurier I, Merabtene F, Seksik P, Bourrier A, Cosnes J, Ryffel B, Beaugerie L, Launay JM, Langella P, Xavier RJ, Sokol H. CARD9 impacts colitis by altering gut microbiota metabolism of tryptophan into aryl hydrocarbon receptor ligands. Nat Med. 2016 Jun;22(6):598-605. doi: 10.1038/nm.4102. Epub 2016 May 9. PMID 27158904
- [Background] Le Chatelier E, Nielsen T, Qin J, Prifti E, Hildebrand F, Falony G, Almeida M, Arumugam M, Batto JM, Kennedy S, Leonard P, Li J, Burgdorf K, Grarup N, Jorgensen T, Brandslund I, Nielsen HB, Juncker AS, Bertalan M, Levenez F, Pons N, Rasmussen S, Sunagawa S, Tap J, Tims S, Zoetendal EG, Brunak S, Clement K, Dore J, Kleerebezem M, Kristiansen K, Renault P, Sicheritz-Ponten T, de Vos WM, Zucker JD, Raes J, Hansen T; MetaHIT consortium; Bork P, Wang J, Ehrlich SD, Pedersen O. Richness of human gut microbiome correlates with metabolic markers. Nature. 2013 Aug 29;500(7464):541-6. doi: 10.1038/nature12506. PMID 23985870
- [Background] Lee CH, Steiner T, Petrof EO, Smieja M, Roscoe D, Nematallah A, Weese JS, Collins S, Moayyedi P, Crowther M, Ropeleski MJ, Jayaratne P, Higgins D, Li Y, Rau NV, Kim PT. Frozen vs Fresh Fecal Microbiota Transplantation and Clinical Resolution of Diarrhea in Patients With Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2016 Jan 12;315(2):142-9. doi: 10.1001/jama.2015.18098. PMID 26757463
- [Background] Lennard-Jones JE. Classification of inflammatory bowel disease. Scand J Gastroenterol Suppl. 1989;170:2-6; discussion 16-9. doi: 10.3109/00365528909091339. PMID 2617184
- [Background] Manichanh C, Borruel N, Casellas F, Guarner F. The gut microbiota in IBD. Nat Rev Gastroenterol Hepatol. 2012 Oct;9(10):599-608. doi: 10.1038/nrgastro.2012.152. Epub 2012 Aug 21. PMID 22907164
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986
- [Background] Sokol H, Leducq V, Aschard H, Pham HP, Jegou S, Landman C, Cohen D, Liguori G, Bourrier A, Nion-Larmurier I, Cosnes J, Seksik P, Langella P, Skurnik D, Richard ML, Beaugerie L. Fungal microbiota dysbiosis in IBD. Gut. 2017 Jun;66(6):1039-1048. doi: 10.1136/gutjnl-2015-310746. Epub 2016 Feb 3. PMID 26843508
- [Background] Sokol H, Galperine T, Kapel N, Bourlioux P, Seksik P, Barbut F, Scanzi J, Chast F, Batista R, Joly F, Joly AC, Collignon A, Guery B, Beaugerie L; French Group of Faecal microbiota Transplantation (FGFT). Faecal microbiota transplantation in recurrent Clostridium difficile infection: Recommendations from the French Group of Faecal microbiota Transplantation. Dig Liver Dis. 2016 Mar;48(3):242-7. doi: 10.1016/j.dld.2015.08.017. Epub 2015 Sep 7. PMID 26433619
- [Background] Sokol H. Toward Rational Donor Selection in Faecal Microbiota Transplantation for IBD. J Crohns Colitis. 2016 Apr;10(4):375-6. doi: 10.1093/ecco-jcc/jjw005. Epub 2016 Jan 7. No abstract available. PMID 26746170
- [Background] Suskind DL, Singh N, Nielson H, Wahbeh G. Fecal microbial transplant via nasogastric tube for active pediatric ulcerative colitis. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):27-9. doi: 10.1097/MPG.0000000000000544. PMID 25162366
- [Background] Toruner M, Loftus EV Jr, Harmsen WS, Zinsmeister AR, Orenstein R, Sandborn WJ, Colombel JF, Egan LJ. Risk factors for opportunistic infections in patients with inflammatory bowel disease. Gastroenterology. 2008 Apr;134(4):929-36. doi: 10.1053/j.gastro.2008.01.012. Epub 2008 Jan 11. PMID 18294633
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Vermeire S, Joossens M, Verbeke K, Wang J, Machiels K, Sabino J, Ferrante M, Van Assche G, Rutgeerts P, Raes J. Donor Species Richness Determines Faecal Microbiota Transplantation Success in Inflammatory Bowel Disease. J Crohns Colitis. 2016 Apr;10(4):387-94. doi: 10.1093/ecco-jcc/jjv203. Epub 2015 Oct 29. PMID 26519463
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514